CLINICAL TRIAL: NCT03044366
Title: General Anesthesia Management in 15 Preterm Infant Undergoing Diode Laser Photocoagulation for Retinopathy of Prematurity: A Retrospective Study
Brief Title: General Anesthesia Management in 15 Preterm Infant
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ahmet Selim Ozkan, M.D., Inonu University
Other Study IDs: ASOZKAN-1
Record Dates: First submitted 2016-12-01; First posted 2017-02-07 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Anesthesia Management of Premature Infants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Characteristics of Anesthesia management: Evaluate the average value of these data.
  Interventions: Other: general anesthesia management of preterm infants
- Comorbidities: Evaluate the average value of these data.
  Interventions: Other: general anesthesia management of preterm infants

INTERVENTIONS:
Other: general anesthesia management of preterm infants — general anesthesia management of preterm infants

SUMMARY:
Anesthesia management of preterm infants is challenging for the anesthesiologist. Because of rudimentary build, many medical and physical problems have shown in treatment of disease such as complications, airway problems, temperature disregulation and deficient drug metabolism. This retrospective study evaluates the perioperative management and postoperative course in premature infants undergoing diode laser photocoagulation (DLP) for retinopathy of prematurity (ROP).

DETAILED DESCRIPTION:
Participants retrospectively investigate clinical data and anesthesia process of 15 preterm infant from anesthesia charts with ROP who underwent DLP between 2014 and 2016. This presented retrospective study was confirmed by the Institutional Clinical Research Ethics Board. Neonates burns under 30 weeks gestation and low birth weigh under 2000 g were admitted to the study. No infant were excluded from the study. Preterm infants were appreciated before surgery and informed consent was obtained form their parents. We recorded gestational age, American Society of Anesthesiologists (ASA) physical status scores, post-conceptual age, weight at birth and surgery, duration of anesthesia and surgery, blood glucose values at surgery, the management of airway, total hospital stay period, analgesia management, complications and comorbidities. Bradycardia ( <90 beats/mean), desaturation (SpO2 <90%) and arrhythmia were recorded. Electrocardiography (ECG), pulse oximetric saturation (SpO2), end-tidal carbon dioxide pressure, heart rate (HR) and body temperature were monitored in operating room. Topical 0.5% proparacaine eye drops were administered to all infants routinely. Anesthesia was induced with thiopental 6 mg kg-1 and fentanyl 1 µg kg-1 and it was maintained with 50% oxygen 50% air 1%-3% sevoflurane in all cases. Inhaled anesthetic agent was not preferred for induction of anesthesia because of causing hypotension. The premature infants were intubated by same experienced anesthesiologist. In all infants, were intubated the patients without muscle relaxant under spontaneous ventilation. Perioperative complications, blood glucose value, devices in airway management and extubation value were recorded. After surgery, extubation was performed when spontanea ventilation was enough and extubation was recorded. All infants were taken to newborn intensive care unit (NICU). Data are reported as mean ± standard deviation and percentage(%).

ELIGIBILITY:
Inclusion Criteria:

* all preterm infants who was decided to apply ROP

Exclusion Criteria:

* No patient was excluded

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patiens who were operated about retinopathy of premature.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
the management of airway | up to 2 years
  the management of airway
gestational age | up to 2 years
  gestational age
American Society of Anesthesiologists physical status scores | up to 2 years
  American Society of Anesthesiologists physical status scores
post-conceptual age | up to 2 years
  post-conceptual age
weight at birth and surgery | up to 2 years
  weight at birth and surgery
duration of anesthesia and surgery | up to 2 years
  duration of anesthesia and surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University Medical Faculty, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes